CLINICAL TRIAL: NCT00820638
Title: Myomo NeuroRobotic System Home Safety Study For Use by Stroke Survivors for Upper Extremity Rehabilitation in Their Homes
Brief Title: Myomo e100 NeuroRobotic System Home Safety Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Myomo (Industry)
Responsible Party: Richard Hughes, PT, MS, Myomo, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
Keywords: neurorobotics; occupational therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): observational
  Interventions: Device: myomo e100

INTERVENTIONS:
Device: myomo e100 — use of the myomo e100 in home
  Other Names: neurorobotic system

SUMMARY:
Up to 25 subjects will use the Myomoe100 in the home setting under the distant supervision of an occupational therapist. We will look to see if they can perform functional activities safely without adverse events.

DETAILED DESCRIPTION:
Hypothesis Subjects can safely use the Myomo e100 NeuroRobotic System in the home.

Primary Outcome Measures:

1. Safety:

1. Safety of the device will be measured by the number of unanticipated or significant device related adverse events reported over a three week period of time. Minor known risks anticipated from device use are mild muscle soreness and fatigue. These will not be considered adverse events.

   Secondary objectives & outcome measures:

   A series of secondary outcome measures will be taken for the reasons listed below:

   • ROM in the affected arm will be taken at the elbow, specifically elbow extension and flexion
   * MMT will be taken for the bicep and tricep muscles
   * The Chedoke Arm and Hand Activity Inventory (CAHAI) will be administered at the start and end of the study scale to measure changes in functional recovery of the arm and hand. 4 This is a valid, clinically relevant, responsive functional assessment of the recovering paretic upper limb and uses bilateral, real-life items. Successful changes in this test will be defined as a predetermined minimum increase in scores. This inventory will provide two types of information: 1st baseline measures of the severity of the individual's impairment and functional levels. This will help identify which groups of stroke patients are best suited for this product in the home
   * Additionally, since the subjects will be practicing specific tasks on the Chedoke via repetitive task practice it is anticipated that there may be a change in the Chedoke scores at the end of four weeks.
   * Motor Activity Log, a semi-structured interview for hemiparetic stroke patients will be administered at the study start and end, as well as weekly by the therapist during the weekly visits to assess the use of their paretic arm and hand (amount of use [AOU]) and quality of movement [QOM]) during activities of daily living. It is anticipated that the subject will use the device more each week as the subject is more acquainted with the device and as tasks become easier. 5
   * Data will also be captured to determine if subjects are able to be trained to successfully don, doff, and operate the device via passing a competency exam.
   * Pain in the shoulder, arm, and hand areas will be assessed on a VAS (0-10) weekly at the therapist visit. It is not anticipated that there will be an increase in arm pain beyond normal muscle soreness related to increase utilization of muscle fibers after several months of inactivity.6
   * Skin areas on the affected arm will be examined by the therapist at the weekly visit and noted for redness or skin breakdown.

   Subject Population:

   Goal: 6 (completers) subjects

   (Goal 15 enrolled to accommodate drop outs and those who may not pass the competency exam)

   Study Intervention:

   Initial training:

   Subjects will come to the clinic over a period of 5 days, for up to three, 2 hour sessions each to perform all pre tests, learn how to properly don, operate the device, and to safely perform a series of home activities. The teaching therapist will determine the appropriate device settings for the subject.

   During the first session the subject will:

   1. Review and sign the informed consent form 2. Perform all pre and post tests under the supervision of a therapist 3. Receive an introduction to the device that will include fitting, basic operation and safety related items to operating the device (i.e.) and simple flexion and extension tasks.

   4. The subject will be given a user manual and MAL. He/she will be asked to fill out the MAL so the therapist can get an idea of what the person can do on a daily basis. The subject will be asked to be familiar with the user manual. The subject will return in 2 days.

   During the second training session the subject and therapist will:

   1. Review donning and doffing the brace 2. Review turning the device on and off 3. Review safety and the user manual 4. Take a device competency test to ensure the subject is aware of all safety precautions and basic device operation. If they fail they will be allowed to come back to Myomo for up to 4 additional visit in order to provide an opportunity to pass the competency. .

   5. Next the therapist will program the device specifically to the subject's level of competency. The subject will be given specific device settings based on their ability to perform the tasks in table 1 which the therapist feels is the most appropriate for the patient. The goal of the setting is to provide the subject with assistance with the activities.

   6. The subject will be instructed in how to fill out the home user log. 7. The subject will be provided with the therapist's direct number if any questions related to operation arise.

   The third through sixth visit will be utilized if the subject requires further instruction and review.

   Initial assessments:

   On the first training session, the treating therapist will adminster commonly utilized, non invasive, therapeutic outcome measures. These measures will include but are not limited to: the subject's range of motion( elbow flexion and extension), manual muscle strength in the bicep and tricep, functional measures such as: Chedoke Arm and Hand Activity Inventory (CAHAI), the Motor Activity Log (MAL) and affected arm pain assessment using the Visual Ananlog Scale.(VAS)

   Assigned treatment tasks:

   During 15 sessions, over a period of three weeks, the subjects will then be asked to perform tasks at home with the device on. The subjects will be asked to perform these tasks at home for approximately one hour each session. The frequency of sessions will be: 5 times per week..

   After a brief stretching and warm up period, each subject will be asked to perform muscular re-education and ROM activities. A sample of possible activities put together by a panel of expert therapists can be found in table 1.

   Table 1. # Task Device mode to be used Number of Sets/Reps
   1. Bend and straighten the elbow while seated (bicep/tricep mode) 3sets/10 reps
   2. Straighten the elbow and hold 10 seconds while seated (tricep mode) 3 sets/10 reps
   3. Wall Push Ups/Seated or standing (tricep mode) 3 sets/10 reps
   4. Bicep curls with a rolling pin (bicep mode) 3 sets/10 reps
   5. Pick up a box from various heights (bicep mode) 3 sets/10 reps
   6. Place container on table (focus on straightening the arm) (tricep mode) 3 stes/10 reps
   7. Steady oneself on a counter top while standing x 20 seconds (tricep mode) 3 sets/10 reps
   8. Carry an object in hand from place to place (bicep mode) 3 sets/10 reps
   9. Toss a ball (overhand or underhand) (bicep mode/tricep mode) 3 sets/10 reps
   10. Pick up tooth-brush and brush teeth (bicep mode) 3 sets/10 reps
   11. Pick up glass (bicep mode) 3 sets/10 reps

   The therapist will provide the patient with a work sheet that lists the exercises chosen from the list above, the mode and settings for the device and the number of sets and reps that should be performed.

   Then, after each session the subject will be asked to complete a simple log that tracks compliance.

   If any type of injury occurs when using the device it will be reported by the subject immediately to the therapist or PI via phone. The incident will be thoroughly documented using guidelines set in place by the New England IRB.

   Weekly therapist visit The patient will return to the research laboratory once a week at Myomo,Inc. The therapist will then review the home use journal with the subject and confirm if no adverse events were reported that none occurred.

   Final study visit:

   The last study visit will include post evaluation report. The research therapist will take ROM, MMT measurements, administer the MAL,the CAHAI and the VAS for pain. Finally, a simple questionnaire about the ease of use of the device and satisfaction with use. Any adverse events since the last visit will be recorded.

   Physician visit:

   Any patient who reports upper limb pain, rash, joint swelling, skin changes or skin injury or any other condition associated with use of the device will be directly referred to their treating physician by the PI or study therapist via phone and a follow up letter.

   Adverse Event:

   An Adverse Event is defined as any injury sustained by the subject during the study visits. Examples of occurrences that would be considered Adverse Events include but are not limited to:
   * Bruising of arm soft tissue
   * Spasms
   * Shoulder pain

   All Adverse Events must be noted in the CRF by marking the Adverse Event check box and then providing a detailed description of the Adverse Event in the notes section of the form. In addition to the standard information captured in the CRF, the notes on the Adverse Event should include information about the specific activity (functional, exercise, or otherwise) that the subject was engaged with at the time of the event, as well any relevant circumstances surrounding the event. Any adverse event must be reviewed by the entire study staff. The adverse event must be reported to the NEIRB in a timely manner and not more than 72 hours after the event.

   Serious adverse events must be reported to the NEIRB as soon as possible, but not more than 24 hours after the event.

ELIGIBILITY:
Inclusion criteria:

* Male or female over the age of 18 who experienced no more than one ischemic or hemorrhagic stroke, at least 6 months ago resulting in hemiparesis in one upper extremity
* Upper extremity Fugl Meyer score >10- - subject must score at least a 10 on the UE FM at the baseline screening appointment only.
* Moderate to Low Tone (Modified Ashworth Score <= 3) If there is too much background contraction in the arm, the system will be unable to pick up voluntary contraction from the background noise, and the brace may not be strong enough to counter the muscle tone. Subject's Modified Ashworth at the screening evaluation score should be < 3
* Considered medically stable- medical conditions that are not under control may affect the subject's ability to participate in treatment sessions safely.
* Able to participate in 17 one hour treatment sessions and willing to complete the evaluations- subjects must be willing to attend all evaluation and treatment sessions
* Score < 3 rating of shoulder pain on the visual analog scale (Appendix N) - subjects must be able to safely tolerate the weight of the brace (about 2 lbs) during treatment sessions.
* Brace fits on arm properly and without discomfort (No red marks or discomfort observed in 10 minutes of use)- subjects need to be able to tolerate sessions with the device
* There is a detectable EMG signal in bicep and tricep and the subject is able to use the brace volitionally- Some voluntary muscle activity must exist for the system to be controlled by the subject due to the non-invasive, surface EMG, sensing methodology.

Exclusion Criteria:

* A current medical history of uncontrolled cardiovascular, or pulmonary disease, or other disease that would preclude involvement in a therapeutic treatment - Subjects must be able to tolerate a 45 minute upper-extremity therapy session in order to participate.
* History of neurological disorder other than stroke- other neurological disorders may affect the upper extremity motor performance of subjects.
* Other significant pain or skin irritation in the upper extremity that would be exacerbated if by the use of the brace - While wearing the brace, the system is pressed close to the upper arm and strapped around it. If the subject suffers from dermal breakdown or other skin conditions that may be aggravated by such a situation, they should not be involved in the study.
* Substantial contracture of elbow - The system cannot work in the presence of reduced range of motion due to contractures. A substantial contracture is defined as greater than 20 degrees of elbow flexion contracture measured at the baseline evaluation.
* Severe sensory loss: Score of 2 on the NIH stroke scale for sensory impairment. The system can work on subjects with sensory loss, however the concern is that a subject with severe sensory loss would not know if the system was applying too much force to the arm or if a strap was too tight and therefore not be able to inform their clinician.
* Use of Botox injections in shoulder, arm or hand for the 3 months prior to study start and throughout the duration of the research study. - the use of Botox may alter the subject's performance on upper extremity motor tasks that are being assessed in the research
* Cognitive or perceptual deficits sufficiently severe enough to interfere with ability to follow instructions- If the subject is unable to understand and follow simple instructions or express if the presence of pain, they should not be included. If the subject scores <69 on the Modified Mini Mental Exam or, if in the opinion of the principle investigator the subject can not safely participate in the study, the subject will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
No reported adverse events | 3 weeks of home use

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hughes, MSPT, Principal Investigator — Myomo
Locations (1):
- Myomo Inc, Charlestown, Massachusetts, United States